CLINICAL TRIAL: NCT01167049
Title: Neoadjuvant Chemotherapy With Xeloda in Combination With Paclitaxel in Gastric Cancer With Liver Metastasis
Brief Title: Xeloda Plus Paclitaxel in Gastric Cancer With Liver Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Ji Jiafu/professor, Beijing Cancer Hosptial
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22199
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Gastric Cancer
Keywords: gastric cancer with liver metastasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAPECITABINE (Experimental): Single arm:
  Capecitabine(Xeloda) 1000 mg/m2 bid, d1-14; q3w; Paclitaxel 80mg/m2 d1,d8; q3w; repeat three cycles (approximately 3- months);
  Interventions: Drug: CAPECITABINE

INTERVENTIONS:
Drug: CAPECITABINE — Capecitabine(Xeloda) 1000 mg/m2 bid, d1-14; q3w; Paclitaxel 80mg/m2 d1,d8; q3w; Repeat three cycles (approximately 3- months);
  Other Names: Xeloda

SUMMARY:
To investigate the efficacy of capecitabine combined with paclitaxel as neoadjuvant chemotherapy for gastric cancer with liver metastasis only

DETAILED DESCRIPTION:
Patients with advanced or metastatic gastric cancer have a poor prognosis. The optimal treatment of gastric cancer with liver metastases without other distant metastases remains a matter for debate and there are few prospective clinical trials to explore this area. The aim of this prospective phase II study is to evaluate the optimal treatment of gastric cancer with liver metastases.

In preclinical xenograft models, capecitabine was highly active against several tumors, including breast, colorectal, gastric, and cervical tumors, and against both 5-FU-sensitive and 5-FU-resistant tumors. Intermittent capecitabine (1250 mg/m2 daily dose for 14 days, followed by a 7-day rest period) was shown to be active as a single agent in previously untreated AGC patients, with a response rate of 28.2% in 39 patients. The combination of capecitabine with other drugs, such as cisplatin, oxaliplatin, epirubicin, and docetaxel, had an objective response rate of 40-68% as first-line treatment in patients with AGC.

In human colon cancer xenograft model, thymidine phosphorylase is upregulated and synergy between paclitaxel and capecitabine has been observed. The activity of capecitabine in patients with breast cancer refractory to paclitaxel and anthracyclines suggests that the combination of capecitabine and paclitaxel may be effective in treating patients with advanced breast cancer. Doses recommended are capecitabine 1650 mg/m2 per day orally for 14 days and paclitaxel 175 mg/m2 i.v. every 3 weeks.

In a phase II trial with 45 patients involved, 2 patients showed complete response and 20 showed partial response making the overall response rate 48.9% (95%CI:30.3-63.5%). There was no neutropaenic fever or treatment-related deaths. That study demonstrated that paclitaxel and capecitabine combination chemotherapy was active and highly tolerable.

The rationale of this study was to find out if outcome could be improved after neoadjuvant chemotherapy with paclitaxel and capecitabine with or without local treatment for patients without other distant metastasis than liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory males or females, aged no less than 18 years.
2. ECOG performance status: 0-1.
3. Histologically confirmed gastric adeno-carcinoma.
4. Radiologically confirmed liver metastasis without other distant metastasis.
5. No serious concomitant medical illnesses
6. Life expectancy more than 3 months
7. Be willing and able to comply with the protocol for the duration of the study
8. No Prior treatment for metastatic disease
9. Give signed informed consent

Exclusion Criteria:

1. not fit for the inclusion criteria
2. not able to comply with the protocol
3. with high risks which may compromise the benefit of proposed regimen
4. Active (significant or uncontrolled) gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response will be evaluated using RECIST criteria. Survival data will be analyzed by Kaplan Meier method. 95% CI will be provided | 3 years from last patient enrolled
  Primary Endpoint is PFS (progression free survival), tumor response will be evaluated using RECIST criteria. Survival data will be analyzed by Kaplan Meier method. 95% CI will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, Post-Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China